CLINICAL TRIAL: NCT01890434
Title: Multicenter Open-label Study to Evaluate Efficacy of Gadobutrol-enhanced Cardiac Magnetic Resonance Imaging (CMRI) for Detection of Significant Coronary Artery Disease (CAD) in Subjects With Known or Suspected CAD by a Blinded Image Analysis
Brief Title: Gadobutrol / Gadavist-enhanced Cardiac Magnetic Resonance Imaging (CMRI) to Detect Coronary Artery Disease (CAD)
Acronym: GadaCAD 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15962; 2013-000066-11 (EudraCT Number)
Record Dates: First submitted 2013-06-27; First posted 2013-07-01 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gadobutrol 0.1 mmol/kg body weight (Experimental): Participants received gadobutrol at the total approved standard dose of 0.1 millimole per kilogram body weight (mmol/kg BW) in 2 separate bolus injections: 0.05 mmol/kg BW at peak pharmacologic stress and 0.05 mmol/kg BW at rest via a power injector.
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Participants received gadobutrol at the total approved standard dose of 0.1 millimole per kilogram body weight (mmol/kg BW) in 2 separate bolus injections: 0.05 mmol/kg BW at peak pharmacologic stress and 0.05 mmol/kg BW at rest via a power injector.

SUMMARY:
Subjects being evaluated for suspected or known Coronary artery Disease (CAD) based on signs and/or symptoms, will be invited to participate in the study. The duration for a subject in the study may range from 2 days to 4-6 weeks. One to four visits to the study doctor will be required.

The primary objective of this study is to demonstrate that sensitivity and specificity of gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) exceed pre-specified minimum performance thresholds of 60% and 55%, respectively, and to show superior sensitivity over unenhanced wall motion CMRI at vasodilator rest/stress for the detection of significant CAD. The CMR images acquired with a uniform imaging acquisition software will be evaluated either against the results from routine clinical Coronary Angiography (CA) or Computed Tomography Angiography (CTA), which are the standard of reference.

CMRI and CA/CTA images will be collected for an independent image review (blinded read).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years
* Subjects with suspected or known CAD based on signs and/or (typical or atypical) chest pain who have routine CA without intervention within plus/minus 4 weeks of gadobutrol-enhanced CMRI or subjects at low risk of CAD with / or scheduled to get a CTA for the purpose of exclusion of CAD within plus/minus 6 weeks of gadobutrol-enhanced CMRI
* Willingness to undergo unenhanced wall motion and gadobutrol-enhanced CMRI at stress/rest and gated single photon emission computed tomography (GSPECT, if GSPECT will be a study procedure)
* Women of childbearing potential (e.g. age < 60y, no history of surgical sterilization or hysterectomy): use of contraception and a negative pregnancy test
* Subjects who are scheduled for / have undergone routine GSPECT or undergo GSPECT as a study procedure at stress and at rest within ± 4 weeks of gadobutrol-enhanced CMRI

Exclusion Criteria:

* Suspected clinical instability or unpredictability of the clinical course during the study period
* Contraindication to the cardiac MRI examination (e.g. inability to hold breath; severe claustrophobia, metallic devices such as pace makers)
* History of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents according to the investigator's assessment / judgment
* Estimated glomerular filtration rate (eGFR) value <30 mL/min/1.73 m^2 derived from a serum / blood creatinine result within 2 weeks prior to gadobutrol injection. Any subject on hemodialysis or peritoneal dialysis is excluded from enrollment.
* Acute renal insufficiency
* Coronary artery bypass grafting (CABG)
* Acute myocardial infarction (< 14 days prior to inclusion), unstable angina / acute coronary syndrome, severe congestive heart failure
* Irregular heart rhythm
* Condition that precludes the safe administration of pharmacological stressor according to the respective approved label such as sinus node disease, 2nd or 3rd degree atrioventricular block, obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2013-08-26 (Actual); Primary Completion 2016-08-06 (Actual); Study Completion 2016-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- United States (14):
  - Tucson, Arizona
  - Los Angeles, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - Bethesda, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Charlottesville, Virginia
- Australia (4):
  - Adelaide, South Australia
  - Perth, Western Australia
  - Chermside
  - North Adelaide
- Canada (2):
  - London, Ontario
  - Montreal, Quebec
- Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 24 centers across 4 countries, between 26 August 2013 (first patient first visit) and 06 August 2016 (last patient last visit).
Pre-assignment Details: Overall, 504 participants signed the informed consent, of which 14 did not finish their baseline visit (7 screening failures, 7 dropouts). A total of 490 participants entered the diagnostic imaging phase, of them 478 participants were treated and entered the follow-up phase.
Period: Overall Study
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Started (Treated with gadobutrol) | 478
Evaluated for Efficacy | 389
Completed (Follow-up (FU) completed) | 458
Not Completed | 20
Not completed — Adverse Event | 8
Not completed — PCI at external hospital | 1
Not completed — Assessment discrepancy | 1
Not completed — CRC didn't contact participant for FU | 1
Not completed — Could not get whole set of images | 1
Not completed — Decline to return for GSPECT | 1
Not completed — GSPECT at rest was not done | 1
Not completed — Participant didn't complete MRI | 1
Not completed — Uncontactable by phone | 1
Not completed — Moved out of position | 1
Not completed — Unable to contact | 1
Not completed — Withdrawal by PI for ICA not performed | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF)
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 478
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 448
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 58
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 81
  White | 322
  More than one race | 3
  Unknown or Not Reported | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 356
  Australia | 71
  Singapore | 31
  Canada | 20
Body weight [Mean (Standard Deviation); unit: kilogram (kg)] | 86.2 (18.6)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.9 (9.7)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.4 (5.5)
Childbearing potential [Count of Participants; unit: Participants] — Population: Number of female participants during baseline in SAF = 177
  Participants
    number analyzed (Participants) | 177
    Yes | 27
    No | 150
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 82.0 (18.73)

OUTCOME MEASURES:

1. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Primary Analysis of Sensitivity Based on Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as quantitative coronary angiography (QCA) stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced cardiac magnetic resonance imaging (CMRI) verified by standard of reference (SoR, coronary angiography [CA] or computed tomography angiography [CTA, only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (full analysis set, included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) with significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 150
Sensitivity %
  Reader 1 | 64.7 [56.5 to 72.3]
  Reader 2 | 56.0 [47.7 to 64.1]
  Reader 3 | 61.3 [53.0 to 69.2]

2. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Sensitivity Based on Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) with significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 105
Sensitivity %
  Reader 1 | 77.1 [67.9 to 84.8]
  Reader 2 | 71.4 [61.8 to 79.8]
  Reader 3 | 76.2 [66.9 to 84.0]

3. Primary Outcome: Absence of Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Primary Analysis of Specificity Based on Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/ (true negative + false positive).
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) without significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 238
Specificity %
  Reader 1 | 85.3 [80.1 to 89.5]
  Reader 2 | 88.7 [83.9 to 92.4]
  Reader 3 | 89.5 [84.9 to 93.1]

4. Primary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Specificity Based on Blinded Readers' Assessment
Description: Blinded readers evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/ (true negative + false positive). This additional secondary analysis of specificity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) without significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR.
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 283
Specificity %
  Reader 1 | 82.0 [77.0 to 86.3]
  Reader 2 | 87.3 [82.8 to 90.9]
  Reader 3 | 86.9 [82.4 to 90.6]

5. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Primary Analysis of Sensitivity Comparison Based on the Blinded Readers' Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by blinded readers' assessment. Significant CAD was defined as QCA stenosis of >=50% for primary analysis, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (included all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) with significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 150
Sensitivity %
  Gadobutrol-enhanced CMRI - Reader 1 | 64.7
  Gadobutrol-enhanced CMRI - Reader 2 | 56.0
  Gadobutrol-enhanced CMRI - Reader 3 | 61.3
  Unenhanced CMRI - Reader 1 | 48.0
  Unenhanced CMRI - Reader 2 | 30.0
  Unenhanced CMRI - Reader 3 | 29.3
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 1; Test type: Superiority; p = 0.00009, McNemar; McNemar one-sided test at alpha level of 5%; Sensitivity Difference = 16.7, 95% CI 1-sided [lower limit 9.3]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 2; Test type: Superiority; p < 0.0001, McNemar; McNemar one-sided test at alpha level of 5%; Sensitivity Difference = 26.0, 95% CI 1-sided [lower limit 18.2]
Statistical Analysis 3: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 3; Test type: Superiority; p < 0.0001, McNemar; McNemar one-sided test at alpha level of 5%; Sensitivity Difference = 32.0, 95% CI 1-sided [lower limit 24.5]

6. Primary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Additional Secondary Analysis of Sensitivity Comparison Based on the Blinded Readers' Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by blinded readers' assessment. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 2
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 105
Sensitivity %
  Gadobutrol-enhanced CMRI - Reader 1 | 77.1
  Gadobutrol-enhanced CMRI - Reader 2 | 71.4
  Gadobutrol-enhanced CMRI - Reader 3 | 76.2
  Unenhanced CMRI - Reader 1 | 56.2
  Unenhanced CMRI - Reader 2 | 35.2
  Unenhanced CMRI - Reader 3 | 35.2
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 1; Test type: Superiority; p = 0.00005, McNemar; McNemar one-sided test at alpha level of 2.5%; Sensitivity Difference = 21.0, 95% CI 1-sided [lower limit 12.1]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 2; Test type: Superiority; p < 0.0001, McNemar; McNemar one-sided test at alpha level of 2.5%; Sensitivity Difference = 36.2, 95% CI 1-sided [lower limit 26.3]
Statistical Analysis 3: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI evaluated by Reader 3; Test type: Superiority; p < 0.0001, McNemar; McNemar one-sided test at alpha level of 2.5%; Sensitivity Difference = 41.0, 95% CI 1-sided [lower limit 31.8]

7. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Secondary Analysis of Sensitivity Based on Investigator's Assessment
Description: The investigator evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=50%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 150
Sensitivity % | 72.0 [64.1 to 79.0]

8. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Sensitivity Based on Investigator's Assessment
Description: The investigator evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 105
Sensitivity % | 85.7 [77.5 to 91.8]

9. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Secondary Analysis of Specificity Based on Investigator's Assessment
Description: The investigator evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=50%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/ (true negative + false positive).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 239
Specificity % | 85.8 [80.7 to 89.9]

10. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Specificity Based on Investigator's Assessment
Description: The investigator evaluated 6 myocardial regions based on regional perfusion score [RPS: 0=normal; 1=abnormal, reversible perfusion defect (stress); 2=abnormal, mixed perfusion defect (reversible and fixed/permanent components); 3=abnormal, fixed/permanent perfusion defect/scar (stress and rest)]. A myocardial region was rated to have a perfusion defect in case of a RPS of >=1 and was rated to have normal perfusion in case of a RPS of 0. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/ (true negative + false positive). This additional secondary analysis of specificity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 284
Specificity % | 81.7 [76.7 to 86.0]

11. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus Unenhanced Wall Motion CMRI Images - Secondary Analysis of Sensitivity Comparison Based on the Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by investigator's assessment. Significant CAD was defined as QCA stenosis of >=50%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 5
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 150
Sensitivity %
  Gadobutrol-enhanced CMRI | 72.0
  Unenhanced CMRI | 50.7
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of unenhanced CMRI; Test type: Superiority; p < 0.0001, McNemar; McNemar 2-sided test at alpha level of 5%; Sensitivity Difference = 21.3, 95% CI 2-sided [12.9 to 28.4]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Test type: Superiority; p < 0.0001, McNemar; McNemar 2-sided test at alpha level of 10%; Sensitivity Difference = 21.3, 90% CI 2-sided [14.2 to 27.2]

12. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI and Unenhanced Wall Motion CMRI Images - Additional Secondary Analysis of Sensitivity Comparison Based on the Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus the presence of wall motion abnormalities on unenhanced CMRI images (based on regional perfusion/regional wall motion score of the 6 myocardial regions) was calculated by investigator's assessment. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or the presence of wall motion abnormalities on unenhanced CMRI images verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 2
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 105
Sensitivity %
  Gadobutrol-enhanced CMRI | 85.7
  Unenhanced CMRI | 61.0

13. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus GSPECT - Secondary Analysis of Sensitivity Comparison Based on Majority Blinded Reader's and Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus GSPECT (based on RPS of the 6 myocardial regions) was calculated by majority blinded reader (BR) and investigator's assessment. Significant CAD was defined as QCA stenosis of >=50%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or GSPECT verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) with significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR and available GSPECT.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 141
Sensitivity %
  Gadobutrol-enhanced CMRI - Majority BR: number analyzed (Participants) | 105
  Gadobutrol-enhanced CMRI - Majority BR | 60.0
  Gadobutrol-enhanced CMRI - Investigator | 72.3
  GSPECT - Majority BR: number analyzed (Participants) | 105
  GSPECT - Majority BR | 54.3
  GSPECT - Investigator | 72.3
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of GSPECT evaluated by majority BR; Test type: Non-Inferiority — A non-inferiority margin was set as 15%; p = 0.2733, McNemar; McNemar 2-sided test at alpha level of 5%; Sensitivity Difference = 5.7, 95% CI 2-sided [-5.4 to 14.9]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Sensitivity of gadobutrol-enhanced CMRI was compared with sensitivity of GSPECT evaluated by investigator; Test type: Non-Inferiority — A non-inferiority margin was set as 15%; p = 1.0000, McNemar; McNemar 2-sided test at alpha level of 5%; Sensitivity Difference = 0.0, 95% CI 2-sided [-8.6 to 7.2]

14. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD Per Participant on Gadobutrol-enhanced CMRI and GSPECT - Additional Secondary Analysis of Sensitivity Based on Majority Blinded Reader's and Investigator's Assessment
Description: Presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus GSPECT (based on RPS of the 6 myocardial regions) was calculated by majority blinded reader and investigator's assessment. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or GSPECT verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis. Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR, for assessment on gadobutrol-enhanced CMRI, and available GSPECT for assessment on GSPECT.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 113
Sensitivity %
  Gadobutrol-enhanced CMRI - Majority BR | 78.8
  Gadobutrol-enhanced CMRI - Investigator | 86.7
  GSPECT - Majority BR: number analyzed (Participants) | 77
  GSPECT - Majority BR | 64.9
  GSPECT - Investigator: number analyzed (Participants) | 106
  GSPECT - Investigator | 83.0

15. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI Versus GSPECT -- Secondary Analysis of Specificity Comparison Based on Majority Blinded Reader's and Investigator's Assessment
Description: Absence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus GSPECT (based on RPS of the 6 myocardial regions) was calculated by majority blinded reader and investigator's assessment. Significant CAD was defined as QCA stenosis of >=50%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or GSPECT verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/(true negative + false positive). Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS (all participants who underwent pharmacologic stress and for whom eCRF entries, adequate image sets for unenhanced and gadobutrol-enhanced CMRI, and the complete image set for the SoR diagnosis were available) without significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR and available GSPECT.
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 231
Specificity %
  Gadobutrol-enhanced CMRI - Majority BR: number analyzed (Participants) | 189
  Gadobutrol-enhanced CMRI - Majority BR | 92.1
  Gadobutrol-enhanced CMRI - Investigator | 85.3
  GSPECT - Majority BR: number analyzed (Participants) | 189
  GSPECT - Majority BR | 81.0
  GSPECT - Investigator | 77.5
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Specificity of gadobutrol-enhanced CMRI was compared with specificity of GSPECT by majority BR; Test type: Non-Inferiority — A non-inferiority margin was set as 15%; p = 0.0010, McNemar; McNemar 2-sided test at alpha level of 5%; Specificity Difference = 11.1, 95% CI 2-sided [4.1 to 17.0]
Statistical Analysis 2: Comparison: Gadobutrol 0.1 mmol/kg Body Weight; Specificity of gadobutrol-enhanced CMRI was compared with specificity of GSPECT by investigator; Test type: Non-Inferiority — A non-inferiority margin was set as 15%; p = 0.0094, McNemar; McNemar 2-sided test at alpha level of 5%; Specificity Difference = 7.8, 95% CI 2-sided [1.6 to 13.2]

16. Secondary Outcome: Absence of a Myocardial Perfusion Defect Excluding Significant CAD Per Participant on Gadobutrol-enhanced CMRI and GSPECT - Additional Secondary Analysis of Specificity Based on Majority Blinded Reader's and Investigator's Assessment
Description: Absence of a myocardial perfusion defect on gadobutrol-enhanced CMRI versus GSPECT (based on RPS of the 6 myocardial regions) was calculated by majority blinded reader and investigator's assessment. Significant CAD was defined as QCA stenosis of >=70%, and was determined based on the presence of a myocardial perfusion defect on gadobutrol-enhanced CMRI or GSPECT verified by SoR (CA or CTA [only if disease can be unequivocally rejected]). Specificity= true negative/(true negative + false positive). This additional secondary analysis of specificity was retrospective analysis. Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 14
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 284
Specificity %
  Gadobutrol-enhanced CMRI - Majority blinded reader: number analyzed (Participants) | 283
  Gadobutrol-enhanced CMRI - Majority blinded reader | 86.6
  Gadobutrol-enhanced CMRI - Investigator | 81.7
  GSPECT - Majority blinded reader: number analyzed (Participants) | 223
  GSPECT - Majority blinded reader | 78.9
  GSPECT - Investigator: number analyzed (Participants) | 273
  GSPECT - Investigator | 73.6

17. Secondary Outcome: Localization of a Myocardial Perfusion Defect to Each Coronary Territory on Gadobutrol-enhanced CMRI - Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessment
Description: Sensitivity was calculated coronary territory based, a coronary territory (left anterior descending artery [LAD] / non-LAD / right coronary artery [RCA] / left circumflex artery [LCX]) was rated positive for significant CAD (significant CAD defined as QCA stenosis of>=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Sensitivity was displayed for all 3 blinded readers, majority blinded reader and the investigator.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR in each coronary territory.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 113
Sensitivity %
  Localization to LAD territory - Reader 1: number analyzed (Participants) | 104
  Localization to LAD territory - Reader 1 | 54.8
  Localization to LAD territory - Reader 2: number analyzed (Participants) | 104
  Localization to LAD territory - Reader 2 | 40.4
  Localization to LAD territory - Reader 3: number analyzed (Participants) | 104
  Localization to LAD territory - Reader 3 | 46.2
  Localization to LAD territory - Majority BR: number analyzed (Participants) | 104
  Localization to LAD territory - Majority BR | 48.1
  Localization to LAD territory - Investigator: number analyzed (Participants) | 104
  Localization to LAD territory - Investigator | 52.9
  Localization to non-LAD territory - Reader 1 | 63.7
  Localization to non-LAD territory - Reader 2 | 54.0
  Localization to non-LAD territory - Reader 3 | 63.7
  Localization to non-LAD territory - Majority BR | 61.1
  Localization to non-LAD territory - Investigator | 67.3
  Localization to RCA territory - Reader 1: number analyzed (Participants) | 80
  Localization to RCA territory - Reader 1 | 56.3
  Localization to RCA territory - Reader 2: number analyzed (Participants) | 80
  Localization to RCA territory - Reader 2 | 56.3
  Localization to RCA territory - Reader 3: number analyzed (Participants) | 80
  Localization to RCA territory - Reader 3 | 60.0
  Localization to RCA territory - Investigator: number analyzed (Participants) | 80
  Localization to RCA territory - Investigator | 68.8
  Localization to LCX territory - Reader 1: number analyzed (Participants) | 82
  Localization to LCX territory - Reader 1 | 57.3
  Localization to LCX territory - Reader 2: number analyzed (Participants) | 82
  Localization to LCX territory - Reader 2 | 31.7
  Localization to LCX territory - Reader 3: number analyzed (Participants) | 82
  Localization to LCX territory - Reader 3 | 53.7
  Localization to LCX territory - Investigator: number analyzed (Participants) | 82
  Localization to LCX territory - Investigator | 48.8

18. Secondary Outcome: Localization of a Myocardial Perfusion Defect to LAD and Non-LAD Territory on GSPECT - Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessment
Description: Sensitivity was calculated coronary territory based, a coronary territory (LAD / non-LAD) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Sensitivity was displayed for all 3 blinded readers, majority blinded reader and the investigator. Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR and available GSPECT in each coronary territory, with either blinded reading or investigator reading performed.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 106
Sensitivity %
  Localization to LAD territory - Reader 8: number analyzed (Participants) | 70
  Localization to LAD territory - Reader 8 | 32.9
  Localization to LAD territory - Reader 9: number analyzed (Participants) | 70
  Localization to LAD territory - Reader 9 | 31.4
  Localization to LAD territory - Reader 10: number analyzed (Participants) | 70
  Localization to LAD territory - Reader 10 | 37.1
  Localization to LAD territory - Majority BR: number analyzed (Participants) | 70
  Localization to LAD territory - Majority BR | 31.4
  Localization to LAD territory - Investigator: number analyzed (Participants) | 98
  Localization to LAD territory - Investigator | 43.9
  Localization to non-LAD territory - Reader 8: number analyzed (Participants) | 81
  Localization to non-LAD territory - Reader 8 | 58.0
  Localization to non-LAD territory - Reader 9: number analyzed (Participants) | 81
  Localization to non-LAD territory - Reader 9 | 45.7
  Localization to non-LAD territory - Reader 10: number analyzed (Participants) | 81
  Localization to non-LAD territory - Reader 10 | 45.7
  Localization to non-LAD territory - Majority BR: number analyzed (Participants) | 81
  Localization to non-LAD territory - Majority BR | 48.1
  Localization to non-LAD territory - Investigator | 64.2

19. Secondary Outcome: Localization of a Myocardial Perfusion Defect to Each Coronary Territory on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessment
Description: Sensitivity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Sensitivity was displayed for all 3 blinded readers and the investigator. This additional secondary analysis of sensitivity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR in each coronary territory, with either blinded reading or investigator reading performed.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 77
Sensitivity %
  Localization to LAD territory - Reader 1: number analyzed (Participants) | 63
  Localization to LAD territory - Reader 1 | 74.6
  Localization to LAD territory - Reader 2: number analyzed (Participants) | 63
  Localization to LAD territory - Reader 2 | 58.7
  Localization to LAD territory - Reader 3: number analyzed (Participants) | 63
  Localization to LAD territory - Reader 3 | 63.5
  Localization to LAD territory - Investigator: number analyzed (Participants) | 63
  Localization to LAD territory - Investigator | 68.3
  Localization to non-LAD territory - Reader 1 | 71.4
  Localization to non-LAD territory - Reader 2 | 68.8
  Localization to non-LAD territory - Reader 3 | 74.0
  Localization to non-LAD territory - Investigator | 81.8
  Localization to RCA territory - Reader 1: number analyzed (Participants) | 59
  Localization to RCA territory - Reader 1 | 69.5
  Localization to RCA territory - Reader 2: number analyzed (Participants) | 59
  Localization to RCA territory - Reader 2 | 71.2
  Localization to RCA territory - Reader 3: number analyzed (Participants) | 59
  Localization to RCA territory - Reader 3 | 71.2
  Localization to RCA territory - Investigator: number analyzed (Participants) | 59
  Localization to RCA territory - Investigator | 79.7
  Localization to LCX territory - Reader 1: number analyzed (Participants) | 48
  Localization to LCX territory - Reader 1 | 68.8
  Localization to LCX territory - Reader 2: number analyzed (Participants) | 48
  Localization to LCX territory - Reader 2 | 43.8
  Localization to LCX territory - Reader 3: number analyzed (Participants) | 48
  Localization to LCX territory - Reader 3 | 75.0
  Localization to LCX territory - Investigator: number analyzed (Participants) | 48
  Localization to LCX territory - Investigator | 66.7

20. Secondary Outcome: Localization of a Myocardial Perfusion Defect to Each Coronary Territory on Gadobutrol-enhanced CMRI - Secondary Analysis of Specificity Based on Blinded Readers' and Investigator's Assessment
Description: Specificity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Specificity was displayed for all 3 blinded readers and the investigator.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS without significant CAD (defined as QCA stenosis of >= 50% by) as verified by SoR in each coronary territory, with either blinded reading or investigator reading performed.
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 302
Specificity %
  Localization to LAD territory - Reader 1: number analyzed (Participants) | 277
  Localization to LAD territory - Reader 1 | 89.9
  Localization to LAD territory - Reader 2: number analyzed (Participants) | 277
  Localization to LAD territory - Reader 2 | 92.4
  Localization to LAD territory - Reader 3: number analyzed (Participants) | 277
  Localization to LAD territory - Reader 3 | 92.4
  Localization to LAD territory - Majority BR: number analyzed (Participants) | 277
  Localization to LAD territory - Majority BR | 92.4
  Localization to LAD territory - Investigator: number analyzed (Participants) | 278
  Localization to LAD territory - Investigator | 89.9
  Localization to non-LAD territory - Reader 1: number analyzed (Participants) | 268
  Localization to non-LAD territory - Reader 1 | 83.6
  Localization to non-LAD territory - Reader 2: number analyzed (Participants) | 268
  Localization to non-LAD territory - Reader 2 | 87.3
  Localization to non-LAD territory - Reader 3: number analyzed (Participants) | 268
  Localization to non-LAD territory - Reader 3 | 87.3
  Localization to non-LAD territory - Majority: number analyzed (Participants) | 268
  Localization to non-LAD territory - Majority | 86.9
  Localization to non-LAD territory - Investigator: number analyzed (Participants) | 269
  Localization to non-LAD territory - Investigator | 84.8
  Localization to RCA territory - Reader 1: number analyzed (Participants) | 301
  Localization to RCA territory - Reader 1 | 84.1
  Localization to RCA territory - Reader 2: number analyzed (Participants) | 301
  Localization to RCA territory - Reader 2 | 86.7
  Localization to RCA territory - Reader 3: number analyzed (Participants) | 301
  Localization to RCA territory - Reader 3 | 86.4
  Localization to RCA territory - Investigator | 86.1
  Localization to LCX territory - Reader 1: number analyzed (Participants) | 299
  Localization to LCX territory - Reader 1 | 86.3
  Localization to LCX territory - Reader 2: number analyzed (Participants) | 299
  Localization to LCX territory - Reader 2 | 92.3
  Localization to LCX territory - Reader 3: number analyzed (Participants) | 299
  Localization to LCX territory - Reader 3 | 87.3
  Localization to LCX territory - Investigator: number analyzed (Participants) | 300
  Localization to LCX territory - Investigator | 89.0

21. Secondary Outcome: Localization of a Myocardial Perfusion Defect to LAD and Non-LAD Territory on GSPECT - Secondary Analysis of Specificity Based on Blinded Readers' and Investigator's Assessment
Description: Specificity was calculated coronary territory based, a coronary territory (LAD / non-LAD) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Specificity was displayed for all 3 blinded readers, majority blinded reader and the investigator. Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS without significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR and available GSPECT in each coronary territory, with either blinded reading or investigator reading,
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 267
Specificity %
  Localization to LAD territory - Reader 8: number analyzed (Participants) | 219
  Localization to LAD territory - Reader 8 | 88.6
  Localization to LAD territory - Reader 9: number analyzed (Participants) | 219
  Localization to LAD territory - Reader 9 | 89.5
  Localization to LAD territory - Reader 10: number analyzed (Participants) | 219
  Localization to LAD territory - Reader 10 | 90.9
  Localization to LAD territory - Majority BR: number analyzed (Participants) | 219
  Localization to LAD territory - Majority BR | 91.8
  Localization to LAD territory - Investigator | 88.0
  Localization to non-LAD territory - Reader 8: number analyzed (Participants) | 208
  Localization to non-LAD territory - Reader 8 | 75.0
  Localization to non-LAD territory - Reader 9: number analyzed (Participants) | 208
  Localization to non-LAD territory - Reader 9 | 85.1
  Localization to non-LAD territory - Reader 10: number analyzed (Participants) | 208
  Localization to non-LAD territory - Reader 10 | 88.0
  Localization to non-LAD territory - Majority BR: number analyzed (Participants) | 208
  Localization to non-LAD territory - Majority BR | 85.6
  Localization to non-LAD territory - Investigator: number analyzed (Participants) | 259
  Localization to non-LAD territory - Investigator | 81.1

22. Secondary Outcome: Localization of a Myocardial Perfusion Defect to Each Coronary Territory on Gadobutrol-enhanced CMRI - Additional Secondary Analysis of Specificity Based on Blinded Readers' and Investigator's Assessment
Description: Specificity was calculated coronary territory based, a coronary territory (LAD / non-LAD / RCA / LCX) was rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%), if >=1 myocardial region within the same coronary territory showed a myocardial perfusion defect with a RPS of >=1. A coronary territory (LAD / non-LAD) was rated negative for significant CAD, if no myocardial region within the respective coronary territory showed a myocardial perfusion defect (RPS 0). Specificity was displayed for all 3 blinded readers and the investigator. This additional secondary analysis of specificity was retrospective analysis.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS without significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR in each coronary territory, with either blinded reading or investigator reading.
Measure: Number; unit: Specificity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 341
Specificity %
  Localization to LAD territory - Reader 1: number analyzed (Participants) | 325
  Localization to LAD territory - Reader 1 | 86.8
  Localization to LAD territory - Reader 2: number analyzed (Participants) | 325
  Localization to LAD territory - Reader 2 | 91.1
  Localization to LAD territory - Reader 3: number analyzed (Participants) | 325
  Localization to LAD territory - Reader 3 | 89.8
  Localization to LAD territory - Investigator: number analyzed (Participants) | 326
  Localization to LAD territory - Investigator | 85.6
  Localization to non-LAD territory - Reader 1: number analyzed (Participants) | 311
  Localization to non-LAD territory - Reader 1 | 79.1
  Localization to non-LAD territory - Reader 2: number analyzed (Participants) | 311
  Localization to non-LAD territory - Reader 2 | 85.5
  Localization to non-LAD territory - Reader 3: number analyzed (Participants) | 311
  Localization to non-LAD territory - Reader 3 | 83.0
  Localization to non-LAD territory - Investigator: number analyzed (Participants) | 312
  Localization to non-LAD territory - Investigator | 80.8
  Localization to RCA territory - Reader 1: number analyzed (Participants) | 329
  Localization to RCA territory - Reader 1 | 83.0
  Localization to RCA territory - Reader 2: number analyzed (Participants) | 329
  Localization to RCA territory - Reader 2 | 86.0
  Localization to RCA territory - Reader 3: number analyzed (Participants) | 329
  Localization to RCA territory - Reader 3 | 84.5
  Localization to RCA territory - Investigator: number analyzed (Participants) | 330
  Localization to RCA territory - Investigator | 83.3
  Localization to LCX territory - Reader 1: number analyzed (Participants) | 340
  Localization to LCX territory - Reader 1 | 82.6
  Localization to LCX territory - Reader 2: number analyzed (Participants) | 340
  Localization to LCX territory - Reader 2 | 91.2
  Localization to LCX territory - Reader 3: number analyzed (Participants) | 340
  Localization to LCX territory - Reader 3 | 85.3
  Localization to LCX territory - Investigator | 86.2

23. Secondary Outcome: Detection of Myocardial Perfusion Defect(s) on Gadobutrol-enhanced CMRI in Participants With Significant LMS Stenosis - Based on Blinded Readers' and Investigator's Assessment
Description: Number of participants with myocardial perfusion defects on gadobutrol-enhanced CMRI was calculated in participants with significant left main stem (LMS) stenosis and the myocardial perfusion defect pattern was described. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%).
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with significant LMS stenosis indicating significant CAD (defined as QCA stenosis of >= 50%) as verified by SoR.
Measure: Count of Participants; unit: Participants
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 7
Participants
  Isolated - Reader 1: number analyzed (Participants) | 2
  Isolated - Reader 1 | 1
  Single vessel - Reader 1: number analyzed (Participants) | 1
  Single vessel - Reader 1 | 1
  2-vessel - Reader 1: number analyzed (Participants) | 2
  2-vessel - Reader 1 | 2
  3-vessel - Reader 1: number analyzed (Participants) | 2
  3-vessel - Reader 1 | 1
  Isolated - Reader 2: number analyzed (Participants) | 2
  Isolated - Reader 2 | 0
  Single vessel - Reader 2: number analyzed (Participants) | 1
  Single vessel - Reader 2 | 1
  2-vessel - Reader 2: number analyzed (Participants) | 2
  2-vessel - Reader 2 | 2
  3-vessel - Reader 2: number analyzed (Participants) | 2
  3-vessel - Reader 2 | 1
  Isolated - Reader 3: number analyzed (Participants) | 2
  Isolated - Reader 3 | 1
  Single vessel - Reader 3: number analyzed (Participants) | 1
  Single vessel - Reader 3 | 1
  2-vessel - Reader 3: number analyzed (Participants) | 2
  2-vessel - Reader 3 | 2
  3-vessel - Reader 3: number analyzed (Participants) | 2
  3-vessel - Reader 3 | 1
  Isolated - Majority BR: number analyzed (Participants) | 2
  Isolated - Majority BR | 1
  Single vessel - Majority BR: number analyzed (Participants) | 1
  Single vessel - Majority BR | 1
  2-vessel - Majority BR: number analyzed (Participants) | 2
  2-vessel - Majority BR | 2
  3-vessel - Majority BR: number analyzed (Participants) | 2
  3-vessel - Majority BR | 1
  Isolated - Investigator: number analyzed (Participants) | 2
  Isolated - Investigator | 2
  Single vessel - Investigator: number analyzed (Participants) | 1
  Single vessel - Investigator | 1
  2-vessel - Investigator: number analyzed (Participants) | 2
  2-vessel - Investigator | 2
  3-vessel - Investigator: number analyzed (Participants) | 2
  3-vessel - Investigator | 2

24. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD in Participants With Single or Multi-vessel Disease Evaluated on Gadobutrol-enhanced CMRI - Secondary Analysis of Sensitivity Based on Blinded Readers' and Investigator's Assessment
Description: Sensitivity was calculated for detection of myocardial perfusion defects on gadobutrol-enhanced CMRI in participants with single and multi-vessel diseases. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=50%). Sensitivity= true positive/ (true positive + false negative).
Time Frame: 0 to 30/40 min post-injection
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 84
Sensitivity %
  Single-vessel - Reader 1: number analyzed (Participants) | 59
  Single-vessel - Reader 1 | 45.8 [32.7 to 59.2]
  Single-vessel - Reader 2: number analyzed (Participants) | 59
  Single-vessel - Reader 2 | 32.2 [20.6 to 45.6]
  Single-vessel - Reader 3: number analyzed (Participants) | 59
  Single-vessel - Reader 3 | 39.0 [26.5 to 52.6]
  Single-vessel - Investigator: number analyzed (Participants) | 59
  Single-vessel - Investigator | 45.8 [32.7 to 59.2]
  Multi-vessel - Reader 1 | 77.4 [67.0 to 85.8]
  Multi-vessel - Reader 2 | 72.6 [61.8 to 81.8]
  Multi-vessel - Reader 3 | 77.4 [67.0 to 85.8]
  Multi-vessel - Investigator | 88.1 [79.2 to 94.1]

25. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD in Participants With Single-vessel Disease Evaluated on Gadobutrol-enhanced CMRI and GSPECT - Additional Secondary Analysis of Sensitivity by Majority Blinded Reader and Investigator
Description: Sensitivity was calculated for detection of myocardial perfusion defects on gadobutrol-enhanced CMRI and GSPECT in participants with single-vessel diseases. If >=1 myocardial region showed a myocardial perfusion defect with a RPS of >=1, participants will be rated positive for significant CAD (significant CAD defined as QCA stenosis of >=70%). Sensitivity= true positive/ (true positive + false negative). This additional secondary analysis of sensitivity was retrospective analysis. Blinded reading of the gadobutrol-enhanced CMRI images and GSPECT images was performed by different readers.
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with single-vessel disease indicating significant CAD (defined as QCA stenosis of >= 70%) as verified by SoR.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 27
Sensitivity %
  Gadobutrol-enhanced CMRI - Majority BR | 66.7
  Gadobutrol-enhanced CMRI - Investigator | 70.4
  GSPECT - Majority BR: number analyzed (Participants) | 19
  GSPECT - Majority BR | 21.1
  GSPECT - Investigator: number analyzed (Participants) | 26
  GSPECT - Investigator | 61.5

26. Secondary Outcome: Presence of a Myocardial Perfusion Defect Indicating Significant CAD in Participants With Multi-vessel Disease Evaluated on Gadobutrol-enhanced CMRI and GSPECT - Additional Secondary Analysis of Sensitivity by Majority Blinded Reader and Investigator
Description: as for outcome 25
Time Frame: 0 to 30/40 min post-injection
Population: Participants in FAS with multi-vessel disease indicating significant CAD (defined as QCA stenosis of >=70%) as verified by SoR.
Measure: Number; unit: Sensitivity %
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 74
Sensitivity %
  Gadobutrol-enhanced CMRI - Majority BR | 81.1
  Gadobutrol-enhanced CMRI - Investigator | 90.5
  GSPECT - Majority BR: number analyzed (Participants) | 49
  GSPECT - Majority BR | 77.6
  GSPECT - Investigator: number analyzed (Participants) | 69
  GSPECT - Investigator | 89.9

27. Secondary Outcome: Number of Participants by Their Lowest Confidence in Diagnosis Obtained on Gadobutrol-enhanced CMRI and Unenhanced Wall Motion CMRI - Based on Blinded Readers' and Investigator's Assessment
Description: Score for confidence in diagnosis (not confident, somewhat confident, and confident) was described descriptively for each of the 6 myocardial regions. The frequency over the worst confidence in diagnosis obtained within a participant was displayed. All these analyses were done separately for gadobutrol-enhanced CMRI and unenhanced wall motion CMRI.
Time Frame: 0 to 30/40 min post-injection
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
Number analyzed (Participants) | 389
Participants
  Gadobutrol-enhanced CMRI - Reader 1: Confident | 310
  Gadobutrol-enhanced CMRI - Reader 1: Somewhat confident | 74
  Gadobutrol-enhanced CMRI - Reader 1: Not confident | 4
  Gadobutrol-enhanced CMRI - Reader 1: Missing | 1
  Gadobutrol-enhanced CMRI - Reader 2: Confident | 300
  Gadobutrol-enhanced CMRI - Reader 2: Somewhat confident | 71
  Gadobutrol-enhanced CMRI - Reader 2: Not confident | 17
  Gadobutrol-enhanced CMRI - Reader 2: Missing | 1
  Gadobutrol-enhanced CMRI - Reader 3: Confident | 186
  Gadobutrol-enhanced CMRI - Reader 3: Somewhat confident | 155
  Gadobutrol-enhanced CMRI - Reader 3: Not confident | 47
  Gadobutrol-enhanced CMRI - Reader 3: Missing | 1
  Gadobutrol-enhanced CMRI - Investigator: Confident | 274
  Gadobutrol-enhanced CMRI - Investigator: Somewhat confident | 98
  Gadobutrol-enhanced CMRI - Investigator: Not confident | 17
  Gadobutrol-enhanced CMRI - Investigator: Missing | 0
  Unenhanced CMRI - Reader 1: Confident | 315
  Unenhanced CMRI - Reader 1: Somewhat confident | 72
  Unenhanced CMRI - Reader 1: Not confident | 1
  Unenhanced CMRI - Reader 1: Missing | 1
  Unenhanced CMRI - Reader 2: Confident | 290
  Unenhanced CMRI - Reader 2: Somewhat confident | 84
  Unenhanced CMRI - Reader 2: Not confident | 14
  Unenhanced CMRI - Reader 2: Missing | 1
  Unenhanced CMRI - Reader 3: Confident | 329
  Unenhanced CMRI - Reader 3: Somewhat confident | 44
  Unenhanced CMRI - Reader 3: Not confident | 15
  Unenhanced CMRI - Reader 3: Missing | 1
  Unenhanced CMRI - Investigator: Confident | 341
  Unenhanced CMRI - Investigator: Somewhat confident | 46
  Unenhanced CMRI - Investigator: Not confident | 2
  Unenhanced CMRI - Investigator: Missing | 0

ADVERSE EVENTS:
Time Frame: From the time of gadobutrol injection until 24 ± 6 hours follow-up
Groups:
- Gadobutrol 0.1 mmol/kg Body Weight: Participants received gadobutrol at the total approved standard dose of 0.1 mmol/kg BW in 2 separate bolus injections: 0.05 mmol/kg BW at peak pharmacologic stress and 0.05 mmol/kg BW at rest via a power injector.
Arm/Group | Gadobutrol 0.1 mmol/kg Body Weight
All-Cause Mortality (participants affected / at risk) | 0/478
Serious Adverse Events (participants affected / at risk) | 4/478
Other Adverse Events (participants affected / at risk) | 79/478
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.1 mmol/kg Body Weight (N=478)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadobutrol 0.1 mmol/kg Body Weight (N=478)
Angina pectoris (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Eye swelling (Eye disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (14)
Tongue ulceration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site pruritus (General disorders) | 1 (1)
Application site rash (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 10 (10)
Chest pain (General disorders) | 5 (5)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Feeling cold (General disorders) | 1 (1)
Feeling hot (General disorders) | 2 (2)
Feeling jittery (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Infusion site extravasation (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 6 (6)
Head discomfort (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 25 (27)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less